CLINICAL TRIAL: NCT01710891
Title: Laryngoscope Versus CMAC for Endotracheal Intubation in Patients Undergoing Emergent Airway Management
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hennepin Healthcare Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSR 11-3338
Record Dates: First submitted 2012-10-15; First posted 2012-10-19 (Estimated); Results first posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2018-12

CONDITIONS: Acute Respiratory Distress
Keywords: endotracheal intubation; direct laryngoscopy; video laryngoscopy
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Direct Laryngoscopy (Active Comparator): Patients will undergo their first intubation attempt with direct laryngoscopy using the CMAC device without video assistance. The video monitor with be covered with a hood.
  Interventions: Procedure: Direct Laryngoscopy
- CMAC (Experimental): Patients will undergo their first intubation attempt using the CMAC videolaryngoscope using video assistance
  Interventions: Procedure: CMAC videolaryngoscope

INTERVENTIONS:
Procedure: CMAC videolaryngoscope — patients are intubated using the CMAC video laryngoscope
  Arms: CMAC
Procedure: Direct Laryngoscopy — Patients undergo their first intubation attempt using direct laryngoscopy with a C-MAC device with the video display covered with a hood.
  Arms: Direct Laryngoscopy

SUMMARY:
Randomized controlled trial of intubation using the C-MAC video laryngoscope versus standard laryngoscopy. Patients who are going to be intubated using standard laryngoscopy will be randomized to have their first intubation attempt done using either standard laryngoscopy or the C-MAC video laryngoscope. Subsequent attempts will be at the discretion of the treating physician.

DETAILED DESCRIPTION:
Experimental Design and Methods:

This will be a prospective randomized controlled trial of intubation using the C-MAC video laryngoscope versus standard laryngoscopy for patients requiring emergent intubation in the Emergency Department.

Study Setting and Population:

This study will be performed at an urban county medical center with approximately 97,000 patient visits per year. Adult patients (age >17) requiring intubation will be enrolled.

Study Protocol:

All ED patients who are unable to adequately breathe on their own requiring emergent intubation for airway management will be screened for inclusion in the study. Identified patients will be deemed eligible when the need for intubation has been determined by the treating physician. Eligible patients will be placed on capnograph, cardiac, blood pressure and pulse oximetry monitors. Patients will be randomly assigned to be intubated using standard laryngoscopy with the C-MAC blade or C-MAC videolaryngoscope. Sealed envelopes containing the randomization assignment for the treatment groups will be kept at the patient's bedside in the stabilization room. Patients will be monitored by oxygen saturation, blood pressure, heart rate, and respiratory rate, which are typical for patients requiring intubation in our ED. Data will be recorded every minute by a trained research assistant at the patient's bedside. The lowest oxygen saturation during the procedure will be recorded for determination of hypoxia. Hypoxia will be defined as an oxygen saturation <93%. The number of attempts made to intubate and the total time to successful intubation will be recorded. An attempt starts when the intubating device enters the patients mouth and ends when the endotracheal tube placement is confirmed or when a new intubating device is put in the patients mouth after the previous device had been removed. Data collection includes the timing and number of breaths given via Bag-Valve-Mask and patient repositioning between the attempts. All treatments will be recorded. Data collection will continue until the patient is discharged from the Emergency Department. The patient's diagnosis at the time of discharge from the ED will be recorded. Patients' charts will be reviewed to determine the diagnosis, occurrence of aspiration pneumonia, ICU length of stay, and inpatient length of stay. Two attempts will be made to contact patients 28 days after study enrollment to determine their condition at that time.

Data Analysis:

Data will be collected by a designated research assistant during the procedure and will then be entered into an EXCEL (Microsoft Corp., Redmond, WA) database for storage. Data will be exported into STATA 10.0 (STATA Corp., College Station, TX) for further analysis. The number of attempts to successful intubation and total time to intubation will be compared using descriptive statistics. Occurrence of hypoxia and aspiration pneumonia will be compared in patients who were intubated with the C-MAC to patients intubated with standard laryngoscopy using Chi-Square tests. Oxygen saturation, ETCO2, and heart rate will be compared in both groups using multiple linear regression.

The length of stay and 28 day follow up between the two groups will be compared using Wilcoxon rank sum tests. In order to detect a 15% difference in the length of stay between the two groups, with a power of 80% and an alpha of 0.05, 100 patients will be required in each group for a total of 200 patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age >17) requiring emergent endotracheal intubation in the Emergency Department using direct laryngoscopy

Exclusion Criteria:

* Physician intends to intubate with a device other than a direct laryngoscope

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2011-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James R Miner, MD, Principal Investigator — Hennepin Healthcare Research Institute
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Driver BE, Prekker ME, Moore JC, Schick AL, Reardon RF, Miner JR. Direct Versus Video Laryngoscopy Using the C-MAC for Tracheal Intubation in the Emergency Department, a Randomized Controlled Trial. Acad Emerg Med. 2016 Apr;23(4):433-9. doi: 10.1111/acem.12933. Epub 2016 Mar 24. PMID 26850232

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Direct Laryngoscopy | CMAC
Started | 95 | 103
Completed | 95 | 103
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Direct Laryngoscopy | CMAC | Total
Number analyzed (Participants) | 95 | 103 | 198
Age, Continuous [Mean (Full Range); unit: years] | 51.6 [19 to 88] | 52.6 [19 to 86] | 52.1 [19 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 41 | 73
  Male | 63 | 62 | 125
Region of Enrollment [Number; unit: participants]
  United States | 95 | 103 | 198

OUTCOME MEASURES:

1. Primary Outcome: First Pass Success in Patients Undergoing Emergency Intubation, Intubated With Either Direct Larynogoscopy or Video Laryngoscopy Using a C-MAC Device.
Description: An attempt is counted as the intubating device entering the patients mouth until it is removed. Intubation success is defined as the endotracheal tube being placed in the patients lungs as confirmed by auscultation and end tidal carbon dioxide
Time Frame: During intubation procedure up to 1 hour
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Direct Laryngoscopy | CMAC
Number analyzed (Participants) | 95 | 103
percentage of participants | 86.3 [79.2 to 93.4] | 92.2 [87.0 to 97.5]

2. Primary Outcome: Time to Intubation
Description: The time in seconds from the time at which the intubating device is first placed in the patient's mouth until the time of successful intubation
Time Frame: From the time the first device entered the patients mouth until successful intubation up to 1 hour
Measure: Mean (95% Confidence Interval); unit: Seconds
Arm/Group | Direct Laryngoscopy | CMAC
Number analyzed (Participants) | 95 | 103
Seconds | 58 [49 to 69] | 61 [46 to 77]

3. Secondary Outcome: Length of Stay
Description: The time in days from hospital admission until discharge.
Time Frame: From the time of hospital admission until discharge up to 28 days
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Direct Laryngoscopy | CMAC
Number analyzed (Participants) | 95 | 103
Days | 9.1 [6.6 to 11.5] | 8.5 [6.6 to 10.3]

4. Secondary Outcome: Aspiration Pneumonia
Description: The occurrence of aspiration pneumonia as defined by the clinical diagnosis in the patients chart and or radiographic determination of aspiration during the 28 days after the intubation procedure
Time Frame: from the time of hospital admission up to 28 days
Measure: Number (95% Confidence Interval); unit: Percentage of Aspiration Pneumonia
Arm/Group | Direct Laryngoscopy | CMAC
Number analyzed (Participants) | 90 | 96
Percentage of Aspiration Pneumonia | 12.2 [5.3 to 19.1] | 7.2 [2.0 to 12.6]

5. Secondary Outcome: Incidence of Hypoxia
Description: Oxygen saturations will be recorded during the procedure, oxygen saturation less than 93% will be considered an occurrence of hypoxia
Time Frame: From the start of the procedure until successful intubation up to 1 hour
Measure: Number (95% Confidence Interval); unit: Percentage of Hypoxemia
Arm/Group | Direct Laryngoscopy | CMAC
Number analyzed (Participants) | 95 | 103
Percentage of Hypoxemia | 27.3 [18.4 to 36.3] | 25.2 [16.9 to 33.6]

6. Secondary Outcome: Failed Intubation
Description: Defined as the operator switching to an alternate device or intubation technique after at least one unsuccessful intubation attempt.
Time Frame: from the start of the procedure until successful intubation up to one hour
Measure: Number; unit: percentage of participants
Arm/Group | Direct Laryngoscopy | CMAC
Number analyzed (Participants) | 13 | 8
percentage of participants | 61.5 | 25

ADVERSE EVENTS:
Arm/Group | Direct Laryngoscopy | CMAC
Serious Adverse Events (participants affected / at risk) | 0/95 | 0/103
Other Adverse Events (participants affected / at risk) | 0/95 | 0/103

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No